CLINICAL TRIAL: NCT02645812
Title: Validation de la Version française du Score de Fatigue " Brief Fatigue Inventory (BFI)
Brief Title: Validation of the French Version of the Fatigue Score "Brief Fatigue Inventory ( BFI)".
Acronym: EAMG
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: EAMG- RB 14.062
Record Dates: First submitted 2016-01-04; First posted 2016-01-05 (Estimated); Last update posted 2016-07-12 (Estimated); Status verified 2016-06

CONDITIONS: Fatigue Symptom
Keywords: Fatigue; Brief Fatigue Inventory (BFI); Primary care; General Practitioners
MeSH Terms: conditions — Fatigue

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Fatigue, or asthenia, is an important symptom for the diagnosis and follow-up of patients in routine as well as research oriented clinical practice.

Various questionnaires measuring fatigue have been developed, but few have been validated in french. MFI (Multidimensional Fatigue Inventory) has been validated in french in only one study. BFI (Brief Fatigue Inventory) has been translated but never validated in french language.

The main purpose of this study is to validate psychometrically the french version of BFI.

ELIGIBILITY:
Inclusion Criteria:

* Consultation for fatigue as symptôme principal ( isolated or asociated with other symptomes).

Exclusion Criteria:

Pregnancy Psychosis. Unable to complete questionnaire Phsyiological fatigue due to effort and reversible rest. Post-traumatic stress disorder -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with fatigue symptom consulting a general practitioner
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2016-03; Primary Completion 2017-09 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
9 points of BFI, each of them between 0 to 10. of BFI | 3 Months

CONTACTS AND LOCATIONS:
Overall Officials: Chritian Berthou, Study Director — CHRU de Brest
Locations (11):
- France (11):
  - Cabinet Brest Centre, Brest
  - Cabinet Camaret/mer, Camaret/mer
  - Cabinet Ergue Gaberic, Ergué-Gabéric
  - Cabinet Le Guilvinec, Guilvinec
  - Cabinet Lamneur, Lanmeur
  - Cabinet Lanmeur, Lanmeur
  - Cabinet Lesconil, Lesconil
  - Cabinet Penmarch, Penmarch
  - Cabinet Plouegat Guerrand, Plouegat Guerrand
  - Cabinet Quimper, Quimper
  - Cabinet Rosporden, Rosporden